CLINICAL TRIAL: NCT03438552
Title: Phase I/II Multi-center Study Evaluating the Efficacy of Repeat Stereotactic Radiation in Patients With Intraprostatic Tumor Recurrence After External Radiation Therapy
Brief Title: Efficacy of Repeat Stereotactic Radiation in Patients With Intraprostatic Tumor Recurrence
Acronym: STEREO-RE-PRO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GETUG-AFU 31 - UC-0160/1618; 2017-A00008-45 (Registry Identifier: ID RCB number)
Record Dates: First submitted 2017-11-14; First posted 2018-02-19 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Local Recurrence of Malignant Tumor of Prostate
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SBRT at a total dose of 30 Gy (Experimental): Placement of fiducials marker seeds in the prostate followed by the administration of stereotactic body radiotherapy at 30 Gy (5 sessions at a level of 6 Gy each- 1 session per day) 30 Gy is the first dose-level. During the treatment phase of the study, no study specific visits are scheduled and the patients will be followed as per standard of care.
  Interventions: Radiation: Stereotactic Body Radiotherapy
- SBRT at a total dose of 25 Gy (Experimental): Placement of fiducials marker seeds in the prostate followed by the administration of stereotactic body radiotherapy at 25 Gy (5 sessions at a level of 5 Gy each- 1 session per day) During the treatment phase of the study, no study specific visits are scheduled and the patients will be followed as per standard of care.
  Interventions: Radiation: Stereotactic Body Radiotherapy
- SBRT at a total dose of 36 Gy (Experimental): Placement of fiducials marker seeds in the prostate followed by the administration of stereotactic body radiotherapy at 36 Gy (6 sessions at a level of 6 Gy each- 1 session per day) During the treatment phase of the study, no study specific visits are scheduled and the patients will be followed as per standard of care.
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — This radiotherapy may be administered with the CyberKnife® or a linear accelerator allowing stereotactic radiotherapy.

SUMMARY:
Stereo-Re-Pro aims to provide further evidence of Stereotactic Body Radiotherapy (SBRT) as a supplementary non-invasive curative treatment for local recurrence following radiotherapy.

The objective of the first part of the trial (Phase I) is to select the recommended dose for salvage SBRT (either 5 x 6 Gy, 6 x 6 Gy, or 5 x 5 Gy) based on dose-limiting toxicity observed during the 18 weeks following the initiation of salvage-SBRT. Particular attention will be paid to the quality of life and tolerance of the treatment.

The objective of the second part of the trial (phase II) is to estimate the efficacy of the salvage-SBRT in terms of biochemical relapse-free survival rate.

DETAILED DESCRIPTION:
To date, no standard local treatment exists for patients with an intraprostatic recurrence after radiotherapy. A number of treatments options exist including: radical prostatectomy, brachytherapy, High-intensity focused ultrasound (HIFU), cryotherapy, and stereotactic radiotherapy. These treatments are associated with a variety of genitourinary and gastrointestinal toxicities and complications. In recent years, stereotactic radiotherapy has been used to treat localized prostate cancer in the primary setting but also as a salvage treatment after failure of radiotherapy. The initial results of these studies are promising, with respect to survival and tolerance, but further studies are required to confirm these initial results.

The objective of STEREO-RE-PRO is to prospectively evaluate salvage SBRT for intraprostatic recurrent prostate cancer after primary external radiotherapy. This study will select patients for whom there is no standard local treatment.

After inclusion and non-inclusion criteria have been verified and the patient has consented, the site will register the screening and organize the baseline visit with the placement of fiducial markers within two months before the planned start of SBRT.

Once the fiducial placement has been performed and all eligibility criteria fully reviewed, the site will register the patient's participation so that the bio-statistician allocates the dose of SBRT. The dose will be allocated upon a model-based estimates provided by the statistical team and confirmed by the trial steering committee. Five or six fractions, at a level of 5 or 6 Gy per session (either 5 x 6 Gy, 6 x 6 Gy, or 5 x 5 Gy), will be delivered over a maximum of 12 days to provide a total dose of 25 to 36 Gy. During the treatment phase of the study, no study specific visits are scheduled and the patients will be followed as per standard of care.

A follow-up visit is planned at 6, 10, 18 weeks from the start of SBRT for safety evaluation. Subsequent follow-up visits are planned at 6, 9, 12, 18, 24, 30, and 36 months after the start of radiotherapy. Thereafter, yearly follow-up visits at 48, 60, and 72 months after starting SBRT will be planned after the initial 3-year follow-up period. M72 visit corresponds to the end of study visit.

ELIGIBILITY:
Inclusion Criteria:

* Biochemical recurrence occurring at least 2 years after external radiotherapy for prostatic adenocarcinoma by the Phoenix definition (PSA nadir + 2 ng/mL)
* T1-T2c and PSA ≤20 ng/mL and Gleason score ≤7 at initial diagnosis of prostate cancer before the initial/first treatment.
* Recurrence of prostatic adenocarcinoma proven by histology following radiotherapy by transrectal or transperineal sextant biopsies of the two lobes of the prostate, with a minimum of 12 biopsies, irrespective of Gleason score. Biopsies of the seminal vesicles are optional.
* Clinical stage T1-T2 on relapse; unilateral extracapsular extension (T3a) on MRI permitted except posteriorly relative to the rectum
* Estimated clinical target volume (CTV) / prostate volume < 0.5 based on imaging and biopsies
* Pelvic and prostatic assessment by multiparametric MRI- Absence of pelvic or metastatic recurrence proven by choline PET scan
* Performance status World Health Organization (WHO) 0-1
* PSA level ≤10 ng/mL at baseline (before salvage-SBRT)
* PSA doubling time >10 months
* International Prostate Cancer Score (IPSS) ≤12
* Uroflowmetry with a maximum flow rate >10 mL/s, a postvoid residual urine volume <150 mL, and a urine volume >150 mL.
* No other anti-cancer treatment since the external radiotherapy administered as first-line treatment
* No other anti-cancer treatment planned for the current recurrence
* No contraindication to fiducial marker implants; haemostatic disorders must be corrected before implantation
* Age >18 years
* Life-expectancy greater than or equal to 5 years (Lee scale)
* Patient registered with a health insurance system
* Patient who has signed the informed consent form
* Patients willing and able to comply with the scheduled visits, treatment plan, laboratory tests, and other study procedures indicated in the protocol.

Exclusion Criteria:

* Lymph node or metastatic spread
* Late post-radiotherapy urinary or gastrointestinal toxicity of grade ≥2 (following primary radiotherapy)
* Other cancers in the last 5 years except for non-melanoma-type skin cancer
* History of inflammatory bowel disease
* Anticoagulant treatment
* Contraindications to undergoing MRI
* Prostate volume >80 cc
* Transurethral resection of the prostate (TURP) in the 6 months before registrations
* Presence of rectal telangiectasia grade 3 classified by the Vienna Rectoscopy Score (obligatory rectoscopy)
* Previous rectal surgery
* Patients unable to undergo medical follow-up in the study for geographical, social or psychological
* Person deprived of their liberty or under protective custody or guardianship
* Patients enrolled in another therapeutic study

All patients during the SBRT planning with a ratio of clinical target volume (CTV) / prostate volume >0.5 will be withdrawn from the study. These patients will be considered as not evaluable and will not be treated within the context of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Selection of the recommended dose for salvage-SBRT (either 5 x 6 Gy, 6 x 6 Gy, or 5 x 5 Gy) based on dose-limiting toxicity observed during the 18 weeks following the initiation of salvage-SBRT. | 18 weeks
  The dose-escalation part of the study will terminate once 10 patients have been treated and evaluated at a dose currently identified as the recommended dose.
Estimate the efficacy of the salvage-SBRT in terms of biochemical relapse-free survival rate | 6 years

SECONDARY OUTCOMES:
Evaluation of acute and late genitourinary toxicities of the salvage-SBRT | 3 years
  Acute and late genitourinary toxicities over the first 3 years according to the NCI-CTCAE V4.03 classification (June 14th, 2010)
Estimate the efficacy of the salvage-SBRT in terms of clinical progression-free survival and overall survival | 6 years
  Clinical progression-free survival is defined as the time interval between the date of registration and the date of clinical progression (local progression assessed by the physical examination, or appearance of metastatic lesions) or death irrespective of the cause.
Evaluation of Quality of life after salvage-SBRT | 6 years
  Quality of life will be evaluated based on the EORTC QLQ-C30. The Time Until Definitive Deterioration (TUDD) will be computed from registration until the first observation of a definitive deterioration of the quality of life, defined as a score decreased by 10 points (in the case of global health scale and functional scales) or increased by 10 points (in the case of symptom scales) compared to the score at baseline, without later improvement superior to 10 points compared to baseline score.
Evaluation of Quality of life after salvage-SBRT | 6 years
  Quality of life will be evaluated based on the EORTC QLQ-PR25. The Time Until Definitive Deterioration (TUDD) will be computed from registration until the first observation of a definitive deterioration of the quality of life, defined as a score decreased by 10 points (in the case of global health scale and functional scales) or increased by 10 points (in the case of symptom scales) compared to the score at baseline, without later improvement superior to 10 points compared to baseline score.

CONTACTS AND LOCATIONS:
Overall Officials: David Pasquier, Principal Investigator — Centre Oscar Lambret, LILLE
Locations (12):
- France (12):
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre George François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut régional du Cancer de Montpellier, Montpellier
  - Groupe Hospitalier Pitié-Salpétrière, Paris
  - DE CREVOISIER Renaud, Rennes
  - ICO -Site René Gauducheau, Saint-Herblain
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - CHRU Henry S.Kaplan, Tours
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pasquier D, Le Deley MC, Tresch E, Cormier L, Duterque M, Nenan S, Lartigau E. GETUG-AFU 31: a phase I/II multicentre study evaluating the safety and efficacy of salvage stereotactic radiation in patients with intraprostatic tumour recurrence after external radiation therapy-study protocol. BMJ Open. 2019 Aug 2;9(8):e026666. doi: 10.1136/bmjopen-2018-026666. PMID 31377694